CLINICAL TRIAL: NCT06521606
Title: Comparison of Temporary External Fixation and Open Reduction With Internal Fixation for the Management of Pilon Fracture: A Prospective Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Omar Sabry, Dr., Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-441-2021
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Pilon Fracture
MeSH Terms: interventions — Fracture Fixation, Internal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- temporary external fixation (Experimental): In our study, 15 patients were managed by the two stages protocol in which they underwent temporary external fixation, and after 7-21 days, they underwent open reduction and internal fixation. The patients were chosen according to the previous criteria; history taking, counselling, general and local examination, and radiological evaluation, and all laboratory investigations were ordered.
  Interventions: Procedure: Temporary external fixator
- Primary open reduction and internal fixation (Active Comparator): Reconstruction and fixation of the metaphyseal shell
  The percutaneous pin was used to manipulate the fragment to achieve reduction; then, a lag screw fixation was done by antegrade technique through a stab incision posteriorly and directly over the fragment. The medial fragment was fixed after the reconstruction of the tibial articular surface to facilitate the anatomic reduction of joint fragments. Again, an image intensifier was used to check the reduction and fixation and to avoid errors of penetration of the joint by screws, malalignment, and inadequate reconstruction of the articular surface; then, the necessary changes were adjusted and made.
  Interventions: Procedure: Primary open reduction and internal fixation

INTERVENTIONS:
Procedure: Primary open reduction and internal fixation — The percutaneous pin was used to manipulate the fragment to achieve reduction; then, a lag screw fixation was done by antegrade technique through a stab incision posteriorly and directly over the fragment. The medial fragment was fixed after the reconstruction of the tibial articular surface to facilitate the anatomic reduction of joint fragments. Again, an image intensifier was used to check the reduction and fixation and to avoid errors of penetration of the joint by screws, malalignment, and inadequate reconstruction of the articular surface; then, the necessary changes were adjusted and made. Wide bone defects in six cases of the primary ORIF cohort and eight cases of the two-stage cohort were packed by corticocancellous iliac bone grafts.
  Arms: Primary open reduction and internal fixation
Procedure: Temporary external fixator — ). Schanz screws with a 6 mm diameter were used to simulate the gripping points on the tibial crest at the proximal metaphyseal or diaphyseal level and on the medial side of the heel bone. This latter pin was carefully inserted medial to lateral, ensuring the starting point is two cm anterior and proximal to the posteroinferior aspect of the calcaneal tuberosity to avoid injury to the medial neurovascular bundle and prevent injury iatrogenic fracture. Such posterior pin placement better balances the deforming forces of the powerful triceps surae muscles. To prevent equinus contracture and provide additional stability. Medial and lateral side rods were then connected to the pins. Manual traction was applied to the exoskeleton base during ligamentotaxis to distract the joint and realign the fracture; this distraction was then kept in place by tightening the clamps.
  Arms: temporary external fixation

SUMMARY:
Pilon fractures are among the difficult injuries to treat in orthopedic surgery. Treatment approaches should consider associated soft tissue injuries. The two main treatment modalities are a two-stage procedure (secondary open reduction internal fixation (ORIF) and primary external fixation) and one-stage ORIF. The latter is widely agreed upon in the literature. In the present study, we contrasted the outcomes of these two approaches.

DETAILED DESCRIPTION:
Pilon fractures are responsible for 1% of lower limb fractures and 5-7% of tibial fractures. The optimal treatment for these fractures has remained challenging and complicated despite significant advancements in recent years in the management of these fractures, mostly because of severely injured soft tissue, severe edema, and a high-energy fracture pattern. As a result, selecting an appropriate course of treatment is still debatable.

Early after the injury, the subcutaneous soft tissue and local skin condition determine whether a direct method and open reconstruction of the articular surface are safe. Early surgical treatment through a flimsy soft tissue envelope raises the possibility of wound complications, promotes infection, and may even result in limb amputation.

The idea of postponing the ultimate osteosynthesis till after the cutaneous condition has been improved came to the forefront in the 1990s. Adopted techniques stressed thorough soft-tissue care in conjunction with delayed definitive fixation to minimize additional damage to surrounding soft tissues. Both long- and short-term outcomes showed decreased surgical complications.

Pilon fractures result from two different force types that can either act individually or concurrently. The primary force is axial compression, resulting in the talus being driven into the tibial plafond; this frequently results in concomitant damage to the talar dome. The secondary force type is rotation, producing variable degrees of articular shearing and fracture fragment displacement. A clear distinction should be made between these two different forces because the relative contribution of each affects the severity of the fracture, soft tissue damage, and prognosis.

The medial fragment, which comprises the medial malleolus and the nearby weight-bearing segment, the Chaput or anterolateral fragment, and the Volkman or posterolateral fragment, typically with their ligamentous attachments intact, are the three variable yet predictable fragments that make up the most specific fracture pattern. Where the implant will be put and, eventually, the surgical approach(es) that will be employed is influenced by the position of the articular segments, the location of the fracture lines as they exit the cortex, and whether or not those parts are continuous with the intact tibial shaft.

The anterolateral quarter of the articular surface and the central corridor of the plafond apex are frequent locations for areas of comminution. As a result, in most patients, an anterior approach provides better access to comminution zones, and an anterolateral distal tibia plate may be employed to strengthen the comminution zone. Although they occur in various planes, the three primary fracture fragments (anterolateral, medial, and posterior) are not sufficiently fixed by a single plate. Most anterolateral plates are insufficiently designed to capture the medial fragment.

Therefore, Phillip Penny et al. stated: Given the wide range of pilon fractures in various patient populations, it is doubtful that a single plate could maintain a sufficient reduction. Hence, it may be best to use a combination of plating techniques to stabilize distal tibia fractures while reinforcing comminution areas.

The results of treating pilon fractures are generally still not satisfactory. Infections, non-union, delayed union, and soft tissue healing complications are common. These complications are mainly caused by the anatomical features of this region, which include limited soft tissue coverage and an insufficient blood supply. Another factor is that such fractures are frequently the result of violent accidents that severely bruise the skin, blood vessels, and muscles. Moreover, in almost two-thirds of cases, arthritis might develop after surgical intervention for pilon fractures.

This study aims to evaluate the feasibility, advantages, and disadvantages of temporary external fixation for pilon fractures and compare its outcomes with cases that will be managed with primary open reduction and internal fixation (ORIF).

ELIGIBILITY:
Inclusion Criteria:

1. Age cohort: adults older than 18 years and less than 70.
2. Sex: both sexes
3. Pilon fracture.

Exclusion Criteria:

1. Patients refused to join the study after explaining the risks and benefits.
2. Infected cases.
3. History of peripheral angiopathy and/or neuropathy in the injured leg.
4. Patients with open fractures.
5. Patients with compartment syndrome.
6. Patients with pathological fractures and associated knee ligament tears.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Primary open reduction and internal fixation | 6 months
  The scale includes nine items that can be divided into three subscales (pain, function and alignment). Pain consists of one item with a maximal score of 40 points, indicating no pain. Function consists of seven items with a maximal score of 50 points, indicating full function. Alignment consists of one item with a maximal score of 10 points, indicating good alignment. The maximal score is 100 points, indicating no symptoms or impairments. In the original publication, the AOFAS Ankle-Hindfoot Score was described to be used for ankle replacement, ankle arthrodesis, ankle instability operations, subtalar arthrodesis, subtalar instability operations, talonavicular arthrodesis, calcaneocuboid arthrodesis, calcaneal osteotomy, calcaneus fracture, talus fracture and ankle fractures

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al Ainy-Cairo University- Faculty of Medicine, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
upon reasonable request.